CLINICAL TRIAL: NCT01577576
Title: Morphological, Biomechanical and Functional Properties of the Arterial Wall of Athletes: Impact and Consequences of Mechanical Stress on the Cardiovascular Adaptations of Peripheral Arterial Calcifications
Brief Title: Mechanical Stress Effects on the Cardiovascular Adaptations of Peripheral Arterial Calcifications Among Athletes
Acronym: MediaSport
Status: Terminated | Type: Observational
Why Stopped: Inclusion curve too slow.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2012/APM-01; 2012-A00475-38 (Other: RCB number)
Record Dates: First submitted 2012-04-12; First posted 2012-04-16 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Monckeberg Medial Calcific Sclerosis
Keywords: Athletes; Sedentary volunteers
MeSH Terms: conditions — Monckeberg Medial Calcific Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — A non-fasting venous blood sample is required for the following cofactors:
  * serum protein
  * serum calcium
  * phosphorus
  * PTH
  * Vitamin D2 and D3
  Left-over serum will be stored in the Nîmes University Hospital "Sérotheque" (serum collection).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Upper-body athletes: This group includes swimmers, rowers or kayakers with a history of at least 10 years of intense training, and performance in regional competitions for the past five years.
- Lower-body athletes: This group includes runners (marathon or trail) and cyclists with a history of at least 10 years of intense training, and performance in regional competitions for the past five years.
- Sedentary volunteers: This group of healthy volunteers does not participate in athletic activity for more than two hours per week. They are matched by age and sex with the athletic groups.

SUMMARY:
The main objective of this study is to obtain data for the integrated analysis of morphological, functional and biomechanical parameters pertaining to lower limb arteries in various categories of elite athletes (without cardiovascular risk and practicing high- or low-impact aerobic activities which preferentially implicate lower limb activity) as compared to (each other and to) sedentary controls.

DETAILED DESCRIPTION:
Secondary objectives of this study are:

A. Determine the presence and extent of intima-media calcifications in athletes B. Determine the relationship between these calcifications and the level, length and intensity of sports activity.

C. Determine the relationship between these properties and calcification of the arterial wall D. Analyze the relationship between the type of sports activity and properties of the arterial wall.

E. Examine the relationship between the properties of the arterial wall and peripheral perfusion pressures.

F. Examine the relationship between the properties of the arterial wall, changes in afterload, morphology and systolic heart function.

G. Analyze the relationships between the parameters characterizing the arterial wall and muscle mass of the lower limbs.

H. Analyze the relationship between the presence of intramural calcification and bone density determined by densitometry.

I. Analyze the relationship between the presence of intramural calcification and dietary protein intake and calcium.

J. Compare indices of pressure at the ankle and toe, depending on the extent of calcification.

K. Create a collection of biological samples (serum).

ELIGIBILITY:
Inclusion Criteria for athletic and sedentary volunteers:

* The volunteer must have given his/her informed and signed consent
* The volunteer must be insured or beneficiary of a health insurance plan
* Volunteers without cardiovascular disease, glucose regulation disorders or known renal disease

Inclusion Criteria for athletic volunteers only:

* Ongoing athletic activity for the past 10 years
* Athletic activity at the regional level for the past 5 years
* Practices one of the three following sports: marathon, trail running, cycling.

Exclusion Criteria for athletic and sedentary volunteers:

* The volunteer is participating in another study
* The volunteer is in an exclusion period determined by a previous study
* The volunteer is under judicial protection, under tutorship or curatorship
* The volunteer refuses to sign the consent
* It is impossible to correctly inform the volunteer
* The volunteer is pregnant, parturient, or breastfeeding
* Tobacco use
* Contraindications for the practice of physical activity (joint, heart or other)
* Intercurrent pathology
* First degree family history of cardiovascular disease
* Known dyslipidemia (including cholesterol)
* Glucose tolerance abnormalities (prediabetes or diabetes)
* Treatment with certain drugs used for treating erectile dysfunction: Sildefanil (Viagra), Tadalafil (Cialis), Vardenafil (Levitra) and yohimbine (Yohimbine Houde and Yocoral)

Exclusion Criteria for sedentary volunteers only:

* More than two hours of athletic activity per week
* History of intense athletic training
* Body mass index >= 25 kg/m^2

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is composed of three groups of healthy volunteers: (1) high impact lower-limb sports (marathon or trail); (2) low-impact lower-limb sports and (3) sedentary volunteers. All volunteers are between the ages of 25 and 40.
  The groups will be matched by age and sex. Athletic groups will be matched according to years of intensive practice and hours of training.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2012-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Presence / absence of intra parietal calcification of lower limb arteries | Baseline (Day 0; transversal study)

SECONDARY OUTCOMES:
Extent of intra parietal calcification of lower limb arteries | Baseline (Day 0; transversal study)
  Score ranging from 0 to 3
Inner diameter of the intima-media of the common femoral artery (mm) | Baseline (Day 0; transversal study)
Outer diameter of the intima-media of the common femoral artery (mm) | Baseline (Day 0; transversal study)
Inner diameter of the intima-media of the superficial femoral artery (mm) | Baseline (Day 0; transversal study)
Outer diameter of the intima-media of the superficial femoral artery (mm) | Baseline (Day 0; transversal study)
Inner diameter of the intima-media of the common carotid artery (mm) | Baseline (Day 0; transversal study)
Outer diameter of the intima-media of the common carotid artery (mm) | Baseline (Day 0; transversal study)
Thickness of the intima-media of the common femoral artery (mm) | Baseline (Day 0; transversal study)
Thickness of the intima-media of the superficial femoral artery (mm) | Baseline (Day 0; transversal study)
Thickness of the intima-media of the common carotid artery (mm) | Baseline (Day 0; transversal study)
Local parietal compliance of the superficial femoral artery | Baseline (Day 0; transversal study)
  mm^2/mmHg
Compliance of the carotid artery | Baseline (Day 0; transversal study)
  mm^2/mmHg
Distensibility of the carotid artery | Baseline (Day 0; transversal study)
  mmHg^-1*10^-2
Arterial wave velocity in lower limb | Baseline (Day 0; transversal study)
  m/s
Arterial wave velocity in upper limb | Baseline (Day 0; transversal study)
  m/s
Endothelium-dependent vasorelaxation in the femoral artery | Baseline (Day 0; transversal study)
Postischemic vasomotor response at the (skin) microcirculatory level | Baseline (Day 0; transversal study)
Systolic pressure index at the ankle | Baseline (Day 0; transversal study)
  relative units
Systolic pressure index for the big toe | Baseline (Day 0; transversal study)
  relative units
Cardiac afterload index | Baseline (Day 0; transversal study)
  g/cm^2
Echocardiographic parameters analyzing systolic function: the stroke volume | Baseline (Day 0; transversal study)
  ml
Echocardiographic parameters analyzing systolic function: cardiac output | Baseline (Day 0; transversal study)
  l/min
Echocardiographic parameters analyzing systolic function: peripheral vascular resistance | Baseline (Day 0; transversal study)
  Pa.s/m^3
Echocardiographic parameters analyzing systolic function: fractional shortening | Baseline (Day 0; transversal study)
Echocardiographic parameters analyzing systolic function: speed of the S-wave according to tissue Doppler | Baseline (Day 0; transversal study)
  cm.s-1
Echocardiographic parameters analyzing systolic function: global longitudinal strain | Baseline (Day 0; transversal study)
Ventricular-arterial coupling | Baseline (Day 0; transversal study)
  relative units
Echocardiographic parameters analyzing diastolic function: transmitral E wave velocity | Baseline (Day 0; transversal study)
  cm/s
Echocardiographic parameters analyzing diastolic function: transmitral A wave velocity | Baseline (Day 0; transversal study)
  cm/s
Echocardiographic parameters analyzing diastolic function: transmitral E wave velocity / transmitral A wave velocity | Baseline (Day 0; transversal study)
  relative units
Echocardiographic parameters analyzing diastolic function: maximum Em wave velocity according to tissue Doppler | Baseline (Day 0; transversal study)
  cm/s
Echocardiographic parameters analyzing diastolic function: maximum Am wave velocity according to tissue Doppler | Baseline (Day 0; transversal study)
  cm/s
Echocardiographic parameters analyzing diastolic function: transmitral E wave velocity / maximum Em wave velocity according to tissue Doppler | Baseline (Day 0; transversal study)
  relative units
Echocardiographic parameters analyzing diastolic function: early diastolic strain-rate | Baseline (Day 0; transversal study)
  s^-1
Years of athletic training | Baseline (Day 0; transversal study)
Hours of athletic training per week | Baseline (Day 0; transversal study)
  h/week
Best performance in the last 6 months | Baseline (Day 0; transversal study)
Lower limb muscle mass | Baseline (Day 0; transversal study)
  g
Bone density | Baseline (Day 0; transversal study)
  g/cm^2
Dietary protein intake | Baseline (Day 0; transversal study)
  g/day
Dietary protein intake | Baseline (Day 0; transversal study)
  % calories per day
Dietary calcium intake | Baseline (Day 0; transversal study)
  mg/day
Serum protein | Baseline (Day 0; transversal study)
  g/l
Serum calcium | Baseline (Day 0; transversal study)
  mmol/l
Serum phosphorus | Baseline (Day 0; transversal study)
  mmol/l
Serum parathyroid hormone | Baseline (Day 0; transversal study)
  ng/l
Serum vitamin D2 | Baseline (Day 0; transversal study)
  µg/l
Serum vitamin D3 | Baseline (Day 0; transversal study)
  µg/l

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Perez Martin, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - Université d'Avignon, Faculté des Sciences, Avignon
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes